CLINICAL TRIAL: NCT06386978
Title: Examination of the Postoperative Analgesic Efficacy of Transvers Abdominis Plane Block and Transversalis Fascia Plane Block in Cesarean Section Surgeries Performed Under Spinal Anesthesia
Brief Title: Analgesic Efficacy of Transvers Abdominis Plane Block and Transversalis Fascia Plane Block in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Kudret Dogru, Prof. Dr., TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/209
Record Dates: First submitted 2024-04-15; First posted 2024-04-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obstetric
Keywords: ceserean section; transverse abdominis plane block; transversalis facia plane block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TAP Group (Active Comparator): TAP (Transverse Abdominis Plane Block) Block was performed in Group 1 patients after negative aspiration on both sides, under aseptic conditions with bupivacaine under ultrasonography guidance.
  Interventions: Procedure: Transverse Facia Plane Block (TAP Block)
- TFP Group (Active Comparator): TFP (Transversalis facia plane block ) Block was performed in Group 2 patients after negative aspiration on both sides, under aseptic conditions with bupivacaine under ultrasonography guidance.
  Interventions: Procedure: Transversalis Facia Plane Block (TFP Block)
- Control Group (Active Comparator): Patients in the Third group will be considered the control group and no block will be performed
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Transverse Facia Plane Block (TAP Block) — Spinal Anesthesia + TAP block
  Arms: TAP Group
Procedure: Transversalis Facia Plane Block (TFP Block) — Spinal Anesthesia + TFP block
  Arms: TFP Group
Procedure: Control — Spinal anesthesia + No block
  Arms: Control Group

SUMMARY:
This study was designed as a prospective, randomized observational clinical trial.

A total of 90 adult women were included in the study performed elective cesarean section.

After excluding patients, the care of 90 was included and 3 of these amounts were reserved.

TAP Block Group (n=30,Group 1): Spinal Anesthesia + TAP block ; TFP Block group (n=30,Group 2): Spinal Anesthesia + TFP block ; Control group (n=30,Group 3); Spinal Anesthesia + No block;

DETAILED DESCRIPTION:
This study was designed as a prospective, randomized observational clinical trial. Erciyes University Clinical Research Ethics Board 2024/209.

All participants in the study were adults and their information was confirmed in writing. Preoperative anesthesia assessment was made by an anesthetic injection, cesarean section surgeries for 90 women were planned to be performed on elective conditions among those registered between May 2024 and May 2025. ASA score, anesthesia method, age, weight, height, TAP block group (Group I) or TFP block group (Group II), Control group (Group III) :

Duration of spinal anesthesia, time of first analgesic request, total analgesic consumption for 24-48 hours, VAS score, additional analgesics, patient satisfaction, possible postoperative bleeding, vomiting, heat retention and other interruptions were recorded in the patients.

Those who were allergic to local anesthetics, steroid treatment areas, ASA III, ASA IV and ASA V, patients under the age of 18, preeclampsia, eclampsia, placenta percreta and accreta complications and emergency hospitals were excluded from the study. After excluding patients, the care of 90 was included and 3 of these amounts were reserved.

TAP Block Group (n=30,Group 1): Spinal Anesthesia + TAP block ; TFP Block group (n=30,Group 2): Spinal Anesthesia + TFP block ; Control group (n=30,Group 3): Spinal Anesthesia + No block; At the end of the surgery, TAP (Transverse Abdominis Plane Block) Block or TFP (Transversalis Fascia Plane Block) block was performed under aseptic conditions under ultrasonography guidance.

TAP (Transverse Abdominis Plane Block) Block for Group 1 patients and TFP (Transversalis Fascia Plane Block) block for Group 2 patients on both sides after negative aspiration, with 20 ml 0.25% bupivacaine (Marcaine®, Astra-Zeneca, Turkey) under ultrasonography guidance. It was done under aseptic conditions.

Patients who did not accept both blocks were included in Group 3 (Control group).

All patients were trained on visual analog score (VAS) by the anesthesia assistant during the preoperative evaluation. VAS used for pain assessment, a 10 cm long horizontal line was used.

From 0= (no pain) to 10= (most severe pain).

PCA morphine administration to all patients: The hourly limit was set as 4 mg, and the repeat limit was set as 10 minutes. If the 1 mg IV morphine bolus dose was not sufficient, it was planned to repeat it after 10 minutes, and if it was still not sufficient, paracetamol and diclofenac were planned to be administered.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and ASA II,
* Pregnant patients accepting spinal anesthesia and procedure

Exclusion Criteria:

* Those who are allergic to local anesthetics,
* Those receiving steroid treatment,
* ASA III, ASA IV and ASA V,
* Patients under the age of 18,
* Patients with preeclampsia,
* Eclampsia,
* Placenta percreta and accreta and its complications,
* Emergency patients.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
VAS score evaluation | 1st, 6th, 12nd, 24 hours at rest, in the first 24hr first day of postoperative period.
  A research asistant, bilinded to the group allocation, interviewedpatients and collected data in the24 hours postoperative period. Verbal Analog Pain Scale Score value will be the lowerst 0 and the highest 10. All the highest value, the patient's pain is at its maximum and whether higher scores mean worse outcome.

SECONDARY OUTCOMES:
time until the first analgesic request | 1st, 6th, 12nd, 24 hours at rest, in the first 24hr first day of postoperative period
  These were the time until the first analgesic request, the number of patients requiring additional analgesics, the general dose of additional analgesic consumption and complications.

OTHER OUTCOMES:
Satisfaction/Dissatisfaction | 1st, 6th, 12nd, 24 hours at rest, in the first 24hr first day of postoperative period
  A scale of Satisfaction/Dissatisfaction was used to evaluate the patient satisfaction rate.

CONTACTS AND LOCATIONS:
Overall Officials: Kudret Dogru, Prof., Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srivastava U, Verma S, Singh TK, Gupta A, Saxsena A, Jagar KD, Gupta M. Efficacy of trans abdominis plane block for post cesarean delivery analgesia: A double-blind, randomized trial. Saudi J Anaesth. 2015 Jul-Sep;9(3):298-302. doi: 10.4103/1658-354X.154732. PMID 26240550
- [Background] Aydin ME, Bedir Z, Yayik AM, Celik EC, Ates I, Ahiskalioglu EO, Ahiskalioglu A. Subarachnoid block and ultrasound-guided transversalis fascia plane block for caesarean section: A randomised, double-blind, placebo-controlled trial. Eur J Anaesthesiol. 2020 Sep;37(9):765-772. doi: 10.1097/EJA.0000000000001222. PMID 32412986